CLINICAL TRIAL: NCT01366053
Title: Hormone Sensitive Prostate Cancer Patients Switched to Degarelix Therapy After Failing on GnRH Agonists: A Prospective, Observational, Phase IV Study (DELAY)
Brief Title: Hormone Sensitive Prostate Cancer Patients Switched to Degarelix Therapy After Failing on GnRH Agonists
Acronym: DELAY
Status: Completed | Type: Observational
Sponsor: CMX Research (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: CMX-DELAY2010
Record Dates: First submitted 2011-05-30; First posted 2011-06-03 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Androgen Deprivation Therapy; Agonist; Antagonist; PSA Failure; PSA Rise
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prostate Cancer: Males who have been diagnosed with Prostate Cancer and are experiencing PSA rise, while taking androgen agonist therapy.

SUMMARY:
This Phase IV observational trial is intended to identify patients who are failing GnRH agonist therapy as evidenced by a rising PSA and who have yet to initiate secondary manoeuvres involving antiandrogens. This group may include both non-metastatic as well as metastatic patients. The trial will determine if these patients will benefit from switching to Degarelix. It will assess the effect of Degarelix's direct mode of action on androgen levels and whether continuous use of Degarelix improves disease progression.

As per the CUA Guidelines for the Management of CRPC, because the androgen receptor remains active in most patients who have developed castration resistant disease, it is recommended that ADT should be continued (LEVEL 3, GRADE C). Therefore, it is logical to continue patients on Degarelix throughout the castrate resistant period. This will allow for the gathering of data that is currently unknown within this setting, such as the effect of combined treatment with antiandrogens as well as chemotherapy and other castrate resistant treatments.

DETAILED DESCRIPTION:
This trial will include hormone sensitive prostate cancer patients switched to Degarelix therapy after failing on GnRH agonists but prior to use of secondary hormonal treatments such as antiandrogens. The purpose of this trial is to determine the effect of Degarelix's direct mode of action on androgen levels and whether continuous use of Degarelix improves disease progression.

This is an open-label, multi-centre, Phase IV observational trial with s.c. injections of Degarelix one-month depot in patients with advanced prostate cancer.

The visit frequency is once a month (28-day intervals), with eCRF data entry at every 4 months. All patients will be treated with a one-month starting dose followed by 23 monthly maintenance doses for a duration of 672 days. The primary endpoints will be evaluated after 24 treatment months.

In total, 25 visits are scheduled for all patients.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and write, understand instructions related to trial procedures and give written informed consent before any trial-related activity is performed
* Histologically confirmed adenocarcinoma of the prostate (prostate cancer)
* Currently under hormonal management of prostate cancer with a GnRH agonist
* Confirmed biochemical PSA progression on GnRH agonist therapy, defined as ≥50% increase in PSA between 2 measurements, taken at least 1 week apart
* PSA ≥1.0 ng/ml
* ECOG score ≤2
* Able and willing to participate in the full duration of the clinical trial
* Male patient aged 18 years or older
* Life expectancy of at least 12 months

Exclusion Criteria:

* Prior treatment with chemotherapy, radiopharmaceuticals, estrogen, ketoconazole or other secondary hormonal treatments such as antiandrogens except for induction phase (<3 months)
* History of dermatitis, lupus, eczema, psoriasis affecting area used for Degarelix injections
* Allergy to Degarelix or its components
* Has a clinically significant disorder (other than prostate cancer) including, but not limited to, renal, haematological, gastrointestinal, endocrine, cardiac, neurological, or psychiatric disease, and alcohol or drug abuse or any other condition, which may affect the patient's health or the outcome of the trial as judged by the Investigator
* Has a history of bilateral orchiectomy, adrenalectomy, or hypophysectomy.
* Has a history of severe untreated asthma, anaphylactic reactions, or severe urticaria and/or angioedema
* Has a mental incapacity or language barrier precluding adequate understanding or co operation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with prostate cancer failing androgen deprivation therapy can be investigated in this trial.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2011-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Testosterone Suppression | Two Years after first dose of degarelix.
  To evaluate testosterone supression in hormone sensitive prostate cancer patients switched to Degarelix therapy after failing on GnRH agonists

SECONDARY OUTCOMES:
Hormone Levels | Two Years after first dose of degarelix.
  To evaluate testosterone, bio available testosterone (calculated), prostate serum antigen (PSA), luteinizing hormone (LH) , follicle-stimulating hormone (FSH), dihydrotestosterone (DHT) and dehydroepiandrosterone (DHEA) before and after switching to Degarelix and over time
PSA Response | Two Years after first dose of degarelix.
  To evaluate PSA response (ability of Degarelix to stabilise or reverse PSA progression)
PSA Failure | Two Years after first dose of degarelix.
  To evaluate how long patients are on degeralix prior to demonstrating biochemical disease progression (time to PSA failure)
PSA Doubling Time | Two Years after first dose of degarelix.
  To evaluate PSA doubling time.
Time to Metastases | Two Years after first dose of degarelix.
  To evaluate how long patients are on degeralix before they develop metastases (non-metastatic patients)
Time to Chemotherapy | Two Years after first dose of degarelix.
  Eevaluate how long patients have been on degeralix before initiating chemotherapy.
Time to Anti-Androgen use | Two Years after first dose of degarelix.
  Evaluate how long patients are on degeralix before initiating anti-androgen use as well as response to anti-androgen use
Patient Performance Status | Two Years after first dose of degarelix.
  To evaluate patient performance status as defined by the Eastern Cooperative Oncology Group (ECOG).

CONTACTS AND LOCATIONS:
Overall Officials: Richard Casey, M.D., Principal Investigator — CMX Research; Alvaro Morales, M.D., Principal Investigator — Queens University
Locations (17):
- Canada (17):
  - Exdeo Clinical Research Inc., Abbotsford, British Columbia
  - Southern Interior Medical Research Inc., Kelowna, British Columbia
  - Andreou Research, Surrey, British Columbia
  - Dr. Steinhoff Clinical Research, Victoria, British Columbia
  - The Male/Female Health and Research Centre, Barrie, Ontario
  - Jonathan Giddens Medicine Professional Corporation, Brampton, Ontario
  - Brantford Urology Research, Brantford, Ontario
  - G. Kenneth Jansz Medicine Professional Corporation, Burlington, Ontario
  - Guelph Urology Associates, Guelph, Ontario
  - Mor Urology Inc., Newmarket, Ontario
  - Toronto Urology Clinical Study Group, North York, Ontario
  - The Fe/Male Health Centres, Oakville, Ontario
  - 2150935 Ontario Inc., Owen Sound, Ontario
  - 643094 Ontario Inc., Scarborough Village, Ontario
  - Stanley Flax Medical Professional Corporation, Toronto, Ontario
  - Urology South Shore Research Inc., Greenfield Park, Quebec
  - Urolaval, Laval, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fontana D, Mari M, Martinelli A, Boccafoschi C, Magno C, Turriziani M, Maymone SS, Cunico SC, Zanollo A, Montagna G, Frongia M, Jacobellis U. 3-month formulation of goserelin acetate ('Zoladex' 10.8-mg depot) in advanced prostate cancer: results from an Italian, open, multicenter trial. Urol Int. 2003;70(4):316-20. doi: 10.1159/000070142. PMID 12740498
- [Background] Gittelman M, Pommerville PJ, Persson BE, Jensen JK, Olesen TK; Degarelix Study Group. A 1-year, open label, randomized phase II dose finding study of degarelix for the treatment of prostate cancer in North America. J Urol. 2008 Nov;180(5):1986-92. doi: 10.1016/j.juro.2008.07.033. Epub 2008 Sep 17. PMID 18801505
- [Background] Jocham D. Leuprorelin three-month depot in the treatment of advanced and metastatic prostate cancer: long-term follow-up results. Urol Int. 1998;60 Suppl 2:18-24; discussion 35. doi: 10.1159/000056547. PMID 9607554
- [Background] Khan MS, O'Brien A. An evaluation of pharmacokinetics and pharmacodynamics of leuprorelin acetate 3M-depot in patients with advanced and metastatic carcinoma of the prostate. Urol Int. 1998;60(1):33-40. doi: 10.1159/000030200. PMID 9519419
- [Background] Morote J, Orsola A, Planas J, Trilla E, Raventos CX, Cecchini L, Catalan R. Redefining clinically significant castration levels in patients with prostate cancer receiving continuous androgen deprivation therapy. J Urol. 2007 Oct;178(4 Pt 1):1290-5. doi: 10.1016/j.juro.2007.05.129. Epub 2007 Aug 14. PMID 17698136
- [Background] Van Poppel H, Tombal B, de la Rosette JJ, Persson BE, Jensen JK, Kold Olesen T. Degarelix: a novel gonadotropin-releasing hormone (GnRH) receptor blocker--results from a 1-yr, multicentre, randomised, phase 2 dosage-finding study in the treatment of prostate cancer. Eur Urol. 2008 Oct;54(4):805-13. doi: 10.1016/j.eururo.2008.04.065. Epub 2008 May 8. PMID 18538469
- [Background] Zinner NR, Bidair M, Centeno A, Tomera K. Similar frequency of testosterone surge after repeat injections of goserelin (Zoladex) 3.6 mg and 10.8 mg: results of a randomized open-label trial. Urology. 2004 Dec;64(6):1177-81. doi: 10.1016/j.urology.2004.07.033. PMID 15596193